CLINICAL TRIAL: NCT03374670
Title: A Phase 2A Open-Label Trial to Assess the Safety of ZIMURA™ (Anti-C5) in Combination With EYLEA® in Treatment Experienced Subjects With Idiopathic Polypoidal Choroidal Vasculopathy
Brief Title: ZIMURA in Combination With Eylea in Patients With Idiopathic Polypoidal Choroidal Vasculopathy (IPCV)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No patients were enrolled. Study terminated for portfolio reasons.
Sponsor: Ophthotech Corporation (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OPH2006
Record Dates: First submitted 2017-12-11; First posted 2017-12-15 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2018-09

CONDITIONS: Idiopathic Polypoidal Choroidal Vasculopathy
Keywords: Zimura; ARC1905; Eylea; aflibercept; IPCV; avacincaptad pegol; complement factor C5 inhibitor
MeSH Terms: conditions — Polypoidal Choroidal Vasculopathy | interventions — aflibercept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): Zimura dosage 1 + Eylea 2 mg
  Interventions: Drug: Zimura; Drug: Eylea
- Cohort 2 (Experimental): Zimura dosage 2 + Eylea 2 mg
  Interventions: Drug: Zimura; Drug: Eylea

INTERVENTIONS:
Drug: Zimura — Zimura in combination with Eylea
  Other Names: avacincaptad pegol
Drug: Eylea — Zimura in combination with Eylea
  Other Names: aflibercept

SUMMARY:
To asses the safety of intravitreal Zimura™ (complement factor C5 inhibitor) administered in combination with Eylea® in treatment experienced subjects with idiopathic polypoidal choroidal vasculopathy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of IPCV
* Patients must have had 3 sequential Eylea injections within the previous 4 months

Exclusion Criteria:

* Intravitreal treatment in the study eye prior to screening, regardless of indication, except 3 prior injections of Eylea
* History or evidence of severe cardiac disease
* Any major surgical procedure within one month of trial entry
* Subjects with a clinically significant laboratory value
* Any treatment with an investigational agent in the past 60 days for any condition
* Women who are pregnant or nursing
* Known serious allergies to the fluorescein dye, ICG dye, iodine, povidone iodine, or to the components or formulation of either Zimura or Eylea

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-11 (Estimated); Primary Completion 2019-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Adverse Events (AEs) | 9 months
  AEs

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Consultants of Hawaii, ‘Aiea, Hawaii, United States